CLINICAL TRIAL: NCT00216021
Title: A Phase II Trial of Capecitabine and Oxaliplatin (CAPOX) in Patients With Metastatic Breast Cancer: Hoosier Oncology Group BRE03-60
Brief Title: Capecitabine and Oxaliplatin in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: Sanofi (Industry); Hoffmann-La Roche (Industry); Walther Cancer Institute (Other)
Responsible Party: Principal Investigator, Kathy Miller, MD, Professor, IU School of Medicine, Hoosier Cancer Research Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOG BRE03-60
Record Dates: First submitted 2005-09-09; First posted 2005-09-22 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Group Assignment (Experimental): Capecitabine + Oxaliplatin
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Capecitabine — Capecitabine 825 mg/m2 po bid, days 1-14
Drug: Oxaliplatin — Oxaliplatin 100 mg/m2 IV, day 1

SUMMARY:
In vitro data suggest synergy between oxaliplatin and 5-FU. The combination of oxaliplatin with 5-fluorouracil produced objective response rates ranging from 27-34% in two studies of patients with prior chemotherapy. Capecitabine was designed as an orally administered, tumor selective fluoropyrimidine, preferentially converted to 5-FU at the tumor site by the higher levels of pyrimidine nucleoside phosphorylase (PyNPase) in tumor tissues compared to normal tissues. The end result is higher concentrations of 5-fluorouracil in tumor relative to surrounding normal tissue. This trial will investigate the activity of this novel capecitabine/oxaliplatin (CAPOX) combination in patients with advanced disease. In addition, an exploratory analysis will correlate response with thymidine synthase and thymidine phosphorylase expression in primary tumor samples.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

CAPOX (21 day cycle):

* Capecitabine 825 mg/m2 orally twice daily Days 1-14.
* Oxaliplatin 100 mg/m2 intravenously Day 1

Patients may continue combination therapy until progression or toxicity intervenes. Patients who discontinue either agent due to toxicity may, at the investigators discretion, continue therapy with the remaining single agent on study.

ECOG performance status 0 or 1

Hematopoietic:·

* ANC > 1,200/mm3·
* Platelets > 100,000/mm3

Hepatic:·

* Total bilirubin < 1.5 x ULN·
* AST < 2 x ULN (up to 5 x ULN in patients with known liver involvement)

Renal:·

* Serum creatinine < 1.5 x ULN and estimated creatinine clearance >50ml/min as calculated with Cockroft-Gault equation

Cardiovascular:·

* No clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of breast cancer with evidence of (1) unresectable, locally recurrent, or (2) metastatic disease.·
* Patients with HER2 positive (3+ overexpression by IHC or gene amplification by FISH) are eligible only if they have had prior trastuzumab therapy.·
* At least one measurable lesion as defined by the RECIST.
* Prior radiation therapy is allowed as long as the irradiated area is not the only source of measurable disease.

Exclusion Criteria:

* No prior therapy with capecitabine or oxaliplatin in any setting
* No prior therapy with other platinum compounds·
* No other forms of cancer therapy including radiation, chemotherapy and hormonal therapy within 21 days prior to beginning protocol therapy.·
* No prior unanticipated severe reaction to fluoropyrimidine therapy, or known sensitivity to 5-fluorouracil.·
* No prior fluoropyrimidine therapy for metastatic disease is allowed. Prior adjuvant fluoropyrimidine therapy is allowed if completed > 12 months from study entry.·
* Maximum of one prior chemotherapy regimen for unresectable, locally recurrent or metastatic disease·
* No symptomatic brain metastasis. ·
* No evidence of serious concomitant systemic disorders incompatible with the study ·
* No peripheral neuropathy ·
* No major surgery within 28 days prior to beginning protocol therapy.·
* Negative pregnancy test·
* No female patients currently breastfeeding·
* No malabsorption syndrome·
* No evidence of serious concomitant systemic disorders incompatible with the study·
* Patients must not be treated with any of the following while on protocol therapy or within 28 days prior to beginning protocol therapy: sorivudine, brivudine, cimetidine, allopurinol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-03; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
- To determine the objective response rate (CR+PR) of capecitabine and oxaliplatin (CAPOX) in patients with metastatic breast cancer. | 36 months

SECONDARY OUTCOMES:
To measure time to progression · | 36 months
To determine rate of clinical benefit response (CR + PR + SD > 6 months). · | 36 months
To determine toxicity rate of CAPOX in this patient population.· | 36 months
To explore potential correlations between thymidine synthase (TS), thymidine phosphorylase (TP) and dihydropyrimidine dehydrogenase (DPD) expression in the primary tumor with response. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Miller, M.D., Study Chair — Hoosier Oncology Group, LLC
Locations (11):
- United States (11):
  - Helen F. Graham Cancer Center, Newark, Delaware
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Oncology Hematology Associates of SW Indiana, Evansville, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Quality Cancer Center (MCGOP), Indianapolis, Indiana
  - Community Regional Cancer Center, Indianapolis, Indiana
  - Medical Consultants, P.C., Muncie, Indiana
  - Center for Cancer Care, Inc., P.C., New Albany, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - AP&S Clinic, Terre Haute, Indiana

REFERENCES:
- See also: Hoosier Oncology Group Home Page — http://www.hoosieroncologygroup.org